CLINICAL TRIAL: NCT07020234
Title: Investigating ELSI Issues That May Facilitate or Impede Clinical Translation of Epigenetic Research: National Survey
Brief Title: National Survey to Understand Ethical, Legal and Social Issues in Communicating to the Public About Epigenetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202503082; R01ES033743 (NIH)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Epigenomics; Epigenetics; Genetics, Behavioral; Bioethics
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epigenetics Video (Experimental): Participants will watch a brief (<5 minute) video about the concept of Epigenetics
  Interventions: Behavioral: Epigenetics Video
- Nanotechnology Video (Active Comparator): Participants will watch a brief (<5 minute) video about nanotechnology
  Interventions: Behavioral: Nanotechnology Video

INTERVENTIONS:
Behavioral: Epigenetics Video — Educational video about health and epigenetics.
  Arms: Epigenetics Video
Behavioral: Nanotechnology Video — Educational video about nanotechnology
  Arms: Nanotechnology Video

SUMMARY:
Few people realize that environmental pollution and some behaviors like physical activity and tobacco smoking can affect their health by "turning on" or "turning off" certain genes through a process called "epigenetic modification." This study will develop and test strategies for communicating about epigenetics that are understandable and that increase acceptance of using epigenetics in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

English language speaker,

Identify as one of five racial/ethnic groups:

1. Non-Hispanic White
2. Non-Hispanic Black,
3. Non-Hispanic Asian
4. Non-Hispanic Indigenous (i.e., Alaska Native/Native Hawaiians/American Indian/Other Pacific Islander)
5. Hispanic (all races)

Exclusion Criteria:

* Self-identify as a genetics expert

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2040 (Actual)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Knowledge & understanding of epigenetics Information | At enrollment
  We will measure this outcome using a sum score of correct answers for 8 individual items.

SECONDARY OUTCOMES:
Acceptability of epigenetics information | At enrollment
  We will measure this outcome using 3 different constructs including perceived benefits of epigenetic research (7 item scale), perceived drawbacks of epigenetic research (3 items), and acceptance of using epigenetic research in medical support (3 items).
Perceptions of epigenetic information | At enrollment
  We will measure this outcome using an 8 item scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT07020234/ICF_000.pdf